CLINICAL TRIAL: NCT05511181
Title: High-frequency Sinusoidal Neurostimulation (BioWave) Versus Transcutaneous Electrical Nerve Stimulation (TENS) for the Treatment of Chronic Low Back Pain
Brief Title: BioWave High-frequency Neurostimulation Versus TENS for the Treatment of Chronic Low Back Pain
Acronym: BioWave
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioWave Corporation (Industry)
Collaborators: Center For Interventional Pain and Spine (Other); Yale University (Other); University of Wisconsin, Madison (Other)
Responsible Party: Principal Investigator, Michael Fishman, MD, Director of Research, Center For Interventional Pain and Spine
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BIOWAVEVSTENSLBP1
Record Dates: First submitted 2022-07-28; First posted 2022-08-22 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Chronic Pain; Lumbar Pain Syndrome; Low Back Pain
Keywords: Chronic Low Back Pain; Lumbar Pain Syndrome
MeSH Terms: conditions — Chronic Pain; Somatoform Disorders; Low Back Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- BioWave (Experimental): BioWaveGO is a FDA 510(k) cleared high frequency neurostimulator. Patients that are first randomized to the BioWave arm will receive a 30 minute treatment in the clinic with a BioWaveGO device followed by a 30 minute washout and ending with a final 30 minute treatment. Data will be collected before, and after the final treatment. Patients will then be instructed to take the BioWaveGO device home and perform two 30 minute treatment sessions daily at home for 2 weeks. Follow-up in the clinic will be after the 2-week treatment period and the patients will be assessed in clinic for physiologic measures of pain response. A washout period of 2 weeks will follow, the patients will return to the clinic at week 4 and the patients will crossover to receive the TENS treatment (as described in the TENS arm).
  Interventions: Device: BioWave
- TENS (Active Comparator): Patients that are first randomized to the TENS arm will receive a 30 minute treatment in the clinic with an Intensity 5000 TENS device followed by a 30 minute washout and ending with a final 30 minute treatment. Data will be collected before, and after the final treatment. Patients will then be instructed to take the TENS device home and perform two 30 minute treatment sessions daily at home for 2 weeks. Follow-up in the clinic will be after the 2-week treatment period and the patients will be assessed in clinic for physiologic measures of pain response. A washout period of 2 weeks will follow, the patients will return to the clinic at week 4 and the patients will crossover to receive the BioWaveGO treatment (as described in the BioWave arm).
  Interventions: Device: TENS

INTERVENTIONS:
Device: BioWave — The BioWave device is called BioWaveGO. It is a FDA 510(k) cleared high frequency sinusoidal neurostimulator
  Arms: BioWave
Device: TENS — The TENS device is called Intensity 5000. It is a FDA 510(k) cleared TENS device
  Arms: TENS

SUMMARY:
This will be a multicenter randomized crossover clinical trial comparing the therapeutic efficacy of BioWave therapy versus TENS for the management of chronic low back pain. This study also aims to evaluate the impact of these therapies on physical activity, patient perception of therapeutic efficacy, and activities of daily living.

DETAILED DESCRIPTION:
This will be a multicenter randomized crossover clinical trial comparing the therapeutic efficacy of BioWave therapy versus TENS for the management of chronic low back pain. This study also aims to evaluate the impact of these therapies on physical activity, patient perception of therapeutic efficacy, and activities of daily living. Patients will start a 30 minute treatment session with either BioWave therapy or TENS device followed by a 30 minute washout and ending with a final 30 minute treatment. Patients will then be instructed to perform two 30 minute treatment sessions daily at home for 2 weeks. Follow-up will be after 2 weeks and the patients will be assessed in clinic for physiologic measures of pain response. A washout period of 2 weeks will follow and the patients will crossover to receive the alternative treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have signed consent before study entry
* Subject must have a body weight of 45 kg or more and a body mass index (BMI) of 40 kg/m2 or less.
* Subject must be aged 18-85 on the date of enrollment and subjects consecutively enrolled
* Subject must have a qualifying baseline pain score of≥5
* Subject must have a stable pain medication regimen for a period of at least 2 weeks prior to study enrollment. Both medication dosages and total number of medications must be stable prior to initiation.
* Subject's pain indication must be defined as chronic low back pain

Exclusion Criteria:

* Subject has a known history of allergic reaction or clinically significant intolerance to medical adhesives, glues, or textiles.
* Subject is currently receiving chronic opioid therapy defined as >30 morphine equivalents units per day (daily use for >2 weeks)
* Subject has an implanted spinal cord stimulator (SCS).
* Subject has any clinically significant clinical, physical, laboratory, or radiographic finding at Screening that, in the opinion of the investigator, contraindicates study participation.
* Subject is currently pregnant.
* Subject has history of or current medical, surgical, post surgical, or psychiatric condition that would confound interpretation of safety, tolerability, or efficacy, (eg, uncontrolled diabetes mellitus, uncontrolled hypertension, hemodynamic instability, or respiratory insufficiency, cancer or palliative care).
* Subject received an experimental drug or used an experimental medical device within 30 days prior to Screening or has previously participated in this trial.
* Subject is unable to comply with the requirements of the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Brief Pain Inventory relative to baseline | completed pre-treatment at the initiation of the study (1st in-clinic treatment), at the 2 week follow up, at week 4, prior to the 2nd in-clinic treatment, and at the 6 week follow up
  Includes a validated short form assessment of pain and function;
  Patient circles the number on a scale of 0 to 10, with 0 meaning no pain and 10 meaning "pain as bad as you can imagine"; a lower score means less pain and a higher score means more pain.
  The higher the score, the worse the outcome.
  Patient circles the one number that describes how, during the past 24 hours, pain has interfered with their life:
  [Scale is between 0-10. 0 means it does not interfere, 10 meaning it completely interferes.
  The higher the score, the worse the outcome.
Change in Visual Analogue Scale relative to baseline | completed pre-treatment and post treatment for the in-clinic visit at week 1 and week 4, as well as at the 2 week and 6 week follow up visits
  straight line with one end meaning no pain and the other end meaning the worst pain imaginable; patient marks a point on the line that matches the amount of pain he or she feels; the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity and a lower score indicates lower pain intensity
Change in Patient Global Impression of Change relative to baseline | completed pre-treatment and post treatment for the in-clinic visit at week 1 and week 4, as well as at the 2 week and 6 week follow up visits
  reflects a patient's belief about the efficacy of treatment; patients will be asked if there overall pain was very much improved, much improved, minimally improved, no change, minimally worse, much worse, or very much worse
Change in Promis-29 relative to baseline | completed pre-treatment at the initiation of the study (1st in-clinic treatment), at the 2 week follow up, at week 4, prior to the 2nd in-clinic treatment, and at the 6 week follow up
  Changes from PROMIS-29 scores relative to baseline for each domain evaluated (physical function, anxiety, depression, fatigue, sleep disturbance, ability to participate in social roles and activities, pain interference, and pain intensity). The first seven domains are assessed with 4 questions each; Pain Intensity is measured with a single 11-point numeric rating scale from 0 (no pain) to 10 (worst imaginable pain). High scores represent more of the domain being measured. On symptom-oriented domains, higher scores signify worse pain. On function-oriented domains, higher scores signify better functioning.

SECONDARY OUTCOMES:
Global assessment of patient impression and perception of pain | completed at the 2 week follow up and the 6 week follow up
  reflects the patient's own assessment of the impact of their condition
  reflects a patient's belief about the efficacy of treatment; patients will be asked if their overall impression and perception of pain was very much improved, much improved, minimally improved, no change, minimally worse, much worse, or very much worse
Global physician assessment of patient improvement | completed at the 2 week follow up and the 6 week follow up
  measures the overall response to treatment as assessed by the physician
  physicians will be asked their overall impression of their patients' improvement was very much improved, much improved, minimally improved, no change, minimally worse, much worse, or very much worse
Change in Blood Pressure (BP) relative to baseline | pre and post at first in-clinic treatment at week 1 and second in-clinic treatment at week 4
  comparison of systolic and diastolic blood pressure measurements
Global assessment of patient impression and perception of quality of life | completed at the 2 week follow up and the 6 week follow up
  reflects the patient's own assessment of their change in quality of life
Change in Heart Rate (HR) relative to baseline | pre and post at first in-clinic treatment at week 1 and second in-clinic treatment at week 4
  comparison of beats per minute
Change in Respiratory Rate (RR) relative to baseline | pre and post at first in-clinic treatment at week 1 and second in-clinic treatment at week 4
  comparison of breaths per minute

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fishman, MD, Principal Investigator — Center For Interventional Pain and Spine
Locations (4):
- United States (4):
  - Yale, New Haven, Connecticut
  - Carolinas Pain Center, Huntersville, North Carolina
  - Center for Interventional Pain and Spine, Lancaster, Pennsylvania
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vance CG, Dailey DL, Rakel BA, Sluka KA. Using TENS for pain control: the state of the evidence. Pain Manag. 2014 May;4(3):197-209. doi: 10.2217/pmt.14.13. PMID 24953072
- [Background] Hegarty DA, Bretherton B. An Open-Label Pilot Study Investigating Noninvasive High-Frequency Peripheral Nerve Fiber Stimulation in Chronic Pain. Pain Pract. 2021 Jun;21(5):578-587. doi: 10.1111/papr.12993. Epub 2021 Jan 27. PMID 33369130
- [Background] S.Diwan, R. F. Eliazo, H. C. Hemmings, S. Panchal: Symptomatic Treatment Of Chronic Low Back Pain: Determination Of Optimal Signal Frequency And Preliminary Efficacy Of A Targeted Non-Invasive Electronic Pain Control Device. Journal of the International Anesthesia Research Society, ANESTH ANALG ABSTRACTS 2003; 96; S-1-S-293
- [Background] Kang RW, Lewis PB, Kramer A, Hayden JK, Cole BJ. Prospective randomized single-blinded controlled clinical trial of percutaneous neuromodulation pain therapy device versus sham for the osteoarthritic knee: a pilot study. Orthopedics. 2007 Jun;30(6):439-45. doi: 10.3928/01477447-20070601-11. No abstract available. PMID 17598487
- [Background] Wanich T, Gelber J, Rodeo S, Windsor R: A Randomized Placebo Controlled Study To Determine Safety and Efficacy In Terms Of Pain Reduction, Increased Range Of Motion, And Reduced Pain Medications, For A Novel Percutaneous Neuromodulation Pain Therapy Device ("Biowave P ENS ®") Following Post - Operative Treatments For Total Knee Replacement Procedures. Poster Presentation American Academy of Orthopaedic Surgeons February 2009
- [Background] Khadilkar A, Odebiyi DO, Brosseau L, Wells GA. Transcutaneous electrical nerve stimulation (TENS) versus placebo for chronic low-back pain. Cochrane Database Syst Rev. 2008 Oct 8;2008(4):CD003008. doi: 10.1002/14651858.CD003008.pub3. PMID 18843638
- [Background] Radhakrishnan R, Sluka KA. Deep tissue afferents, but not cutaneous afferents, mediate transcutaneous electrical nerve stimulation-Induced antihyperalgesia. J Pain. 2005 Oct;6(10):673-80. doi: 10.1016/j.jpain.2005.06.001. PMID 16202960
- [Background] Levin MF, Hui-Chan CW. Conventional and acupuncture-like transcutaneous electrical nerve stimulation excite similar afferent fibers. Arch Phys Med Rehabil. 1993 Jan;74(1):54-60. PMID 8420521
- [Background] Hughes N, Bennett MI, Johnson MI. An investigation into the magnitude of the current window and perception of transcutaneous electrical nerve stimulation (TENS) sensation at various frequencies and body sites in healthy human participants. Clin J Pain. 2013 Feb;29(2):146-53. doi: 10.1097/AJP.0b013e3182579919. PMID 23183261
- [Background] DeSantana JM, Da Silva LF, De Resende MA, Sluka KA. Transcutaneous electrical nerve stimulation at both high and low frequencies activates ventrolateral periaqueductal grey to decrease mechanical hyperalgesia in arthritic rats. Neuroscience. 2009 Nov 10;163(4):1233-41. doi: 10.1016/j.neuroscience.2009.06.056. Epub 2009 Jul 2. PMID 19576962
- [Background] Dailey DL, Rakel BA, Vance CGT, Liebano RE, Amrit AS, Bush HM, Lee KS, Lee JE, Sluka KA. Transcutaneous electrical nerve stimulation reduces pain, fatigue and hyperalgesia while restoring central inhibition in primary fibromyalgia. Pain. 2013 Nov;154(11):2554-2562. doi: 10.1016/j.pain.2013.07.043. Epub 2013 Jul 27. PMID 23900134
- [Background] Hurlow A, Bennett MI, Robb KA, Johnson MI, Simpson KH, Oxberry SG. Transcutaneous electric nerve stimulation (TENS) for cancer pain in adults. Cochrane Database Syst Rev. 2012 Mar 14;2012(3):CD006276. doi: 10.1002/14651858.CD006276.pub3. PMID 22419313
- [Background] Kroeling P, Gross AR, Goldsmith CH; Cervical Overview Group. A Cochrane review of electrotherapy for mechanical neck disorders. Spine (Phila Pa 1976). 2005 Nov 1;30(21):E641-8. doi: 10.1097/01.brs.0000184302.34509.48. PMID 16261102
- [Background] Johnson MI, Mulvey MR, Bagnall AM. Transcutaneous electrical nerve stimulation (TENS) for phantom pain and stump pain following amputation in adults. Cochrane Database Syst Rev. 2015 Aug 18;8(8):CD007264. doi: 10.1002/14651858.CD007264.pub3. PMID 26284511
- [Background] Nnoaham KE, Kumbang J. Transcutaneous electrical nerve stimulation (TENS) for chronic pain. Cochrane Database Syst Rev. 2008 Jul 16;(3):CD003222. doi: 10.1002/14651858.CD003222.pub2. PMID 18646088
- [Background] Rutjes AW, Nuesch E, Sterchi R, Kalichman L, Hendriks E, Osiri M, Brosseau L, Reichenbach S, Juni P. Transcutaneous electrostimulation for osteoarthritis of the knee. Cochrane Database Syst Rev. 2009 Oct 7;2009(4):CD002823. doi: 10.1002/14651858.CD002823.pub2. PMID 19821296
- [Background] Walsh DM, Howe TE, Johnson MI, Sluka KA. Transcutaneous electrical nerve stimulation for acute pain. Cochrane Database Syst Rev. 2009 Apr 15;(2):CD006142. doi: 10.1002/14651858.CD006142.pub2. PMID 19370629